CLINICAL TRIAL: NCT00789698
Title: A Phase 3 Randomized, Double-Blind, Active Comparator-Controlled Clinical Trial to Study the Safety and Efficacy of Lurasidone in Subjects With Schizophrenia (PEARL 3 Extension Study)
Brief Title: Lurasidone HCl - A Long Term Phase 3 Study of Patients With Chronic Schizophrenia
Acronym: PEARL 3 Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1050234
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Schizophrenia
Keywords: Schizophrenia; SM-13496; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lurasidone HC1 (Experimental)
  Interventions: Drug: Lurasidone HC1
- Quetiapine (Active Comparator)
  Interventions: Drug: Quetiapine XR

INTERVENTIONS:
Drug: Lurasidone HC1 — Lurasidone 40-160 mg/day flexibly dosed.
  Arms: Lurasidone HC1
Drug: Quetiapine XR — Quetiapine XR 200-800 mg/day flexibly dosed.
  Arms: Quetiapine

SUMMARY:
Lurasidone HCl is a compound being developed for the treatment of schizophrenia. This clinical study is designed to test the hypothesis that lurasidone is effective, tolerable, and safe as compared with quetiapine XR long term among schizophrenic outpatients with chronic schizophrenia.

ELIGIBILITY:
Entry Criteria:

* Screening for the present study will take place after subjects' participation in Study D1050233 has been completed, and after providing informed consent.

Inclusion Criteria:

* Completed all required assessments on the final study visit in Study D1050233.
* Suitable for treatment in an outpatient setting.

Exclusion Criteria:

* Any chronic organic disease of the CNS (other than schizophrenia).
* Considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (65):
- United States (27):
  - K&S Professional Research Services, LLC, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Comprehensive Neuroscience, Inc, Cerritos, California
  - Clinical Innovations, Inc., Costa Mesa, California
  - Synergy Escondido,710 East Grand Ave., Escondido, California
  - Collaborative Neuroscience Network Inc, Garden Grove, California
  - Apostle Clinical Trials, Inc., Long Beach, California
  - California Clinical Trials, Paramount, California
  - Pasadena Research Institute, Pasadena, California
  - CNRI - Los Angeles LLC,8309 Telegraph Road, Pico Rivera, California
  - CNRI- LOs Angeles, LLC, Pico Rivera, California
  - Clinical Innovations, Inc., Riverside, California
  - CNRI - San Diego, San Diego, California
  - UCSD Medical Drive, Sandeigo, California
  - Segal Institute for Clinical Research, Highlands Ranch, Colorado
  - Comprehensive Neuroscience, Inc., Washington D.C., District of Columbia
  - Florida Clinical Research Center LLC, Bradenton, Florida
  - Lake Charles Clinical Trials LLC,2770 3rd Avenue,Suite 340, Lake Charles, Louisiana
  - Booker, J. Gary, MD. APMC, Shreveport, Louisiana
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - St. Louis Research, Inc., St Louis, Missouri
  - CRI Worldwide, Willingboro, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Comprehensive Neuroscience, Inc, Holliswood, New York
  - Community Clinical Research, Austin, Texas
  - FutureSearch Clinical Trials, LLC., Austin, Texas
  - Pillar Clinical Research, Dallas, Texas
- Colombia (6):
  - CIPNA Centro de Investigaciones y Proyectos en Neurociencias, Calle 80#47-43 Consultorio 5C, Barranquila S/N
  - Centro de Investigacion y Atencion para la Salud Mental, Calle 103A # 21-49, Bogota S/N
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - Centro de Investigación y Atención para la Salud Mental, Bogotá
  - CISNE - UIC Campo Abierto, Bogotá
  - Instituto Colombiano del Sistema Nervioso Clínica Montserrat, Bogotá
- India (10):
  - S.V. Medical College, Tirupati, Andhra Pradesh
  - Vijayawada Institute of Mental Health and Neurosciences, Vijayawada, Andhra Pradesh
  - Shanti Nursing Home, Kanchanpalli, Aurangabad, Maharashtra
  - Seth K M School of P G Medicine & Research, Ahmedabad, Gujarat
  - SBKS Medical College and Hospital, Brij Psychiatry Hospital, Vadodara, Gujarat
  - Justice K.S. Hedge Charitable Hospital, Mangalore, Karna
  - JSS Medical College and Hospital - Dept of Psychiatry, Mysore, Karna
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Mahatma Gandhi Institute of Medical Sciences, Sewāgrām, Maharashtra
  - Madras Medical College & Government General Hospital, Chennai, Tamil Nadu
- Romania (5):
  - Spitalul Clinic Judetean de Urgenta Arad, Str. Octavian Goga Nr. 17, Arad
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Sos. Berceni Nr. 10-12, București
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic de Neurologie si Psihiatrie Oradea, Oradea
  - Spitalul Judetean Arges, Piteşti
- Russia (9):
  - Andreev, Boris, Gatchina
  - Gurovich, Isaak, Moscow
  - Morozova, Margarita, Moscow
  - City Psychoneurological Dispensary #7 (with Hospital), Saint Petersburg
  - City Psyhiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - City Psychiatric Hospital #4, Saint Petersburg
  - City Psychiatric Hospital #3 of Skvortsov-Stepanov, Saint Petersburg
  - Neznanov, Nikolay, Saint Petersburg
  - Sheifer, Mikhail, Samara
- Ukraine (8):
  - Dnipropetrovsk Regional Clinical Hospital named Mechnikov, Dnipropetrovsk
  - Reg.Clin.Psychiatric Hosp., Dept. #11, DSMU n.af.M.Gorkiy, Donetsk
  - Kyiv City Clin. Psychoneurolog. Hosp.#1, Kyiv
  - Kyiv City Psychoneurological Hospital, Kyviv
  - Lviv Reg.St.Cl.Psych.Hosp, Lviv
  - Reg. Psychiatric Hospital, Odesa
  - Crimean republican Clinical Psychiatric Hospital, Simferopol
  - Kherson Regional Psychiatric Hospital, Vil. Stepanovka, Kherson

REFERENCES:
- [Result] Loebel A, Cucchiaro J, Xu J, Sarma K, Pikalov A, Kane JM. Effectiveness of lurasidone vs. quetiapine XR for relapse prevention in schizophrenia: a 12-month, double-blind, noninferiority study. Schizophr Res. 2013 Jun;147(1):95-102. doi: 10.1016/j.schres.2013.03.013. Epub 2013 Apr 11. PMID 23583011
- [Result] Harvey PD, Siu CO, Hsu J, Cucchiaro J, Maruff P, Loebel A. Effect of lurasidone on neurocognitive performance in patients with schizophrenia: a short-term placebo- and active-controlled study followed by a 6-month double-blind extension. Eur Neuropsychopharmacol. 2013 Nov;23(11):1373-82. doi: 10.1016/j.euroneuro.2013.08.003. Epub 2013 Aug 27. PMID 24035633
- [Derived] Harvey PD, Siu CO, Ogasa M, Loebel A. Effect of lurasidone dose on cognition in patients with schizophrenia: post-hoc analysis of a long-term, double-blind continuation study. Schizophr Res. 2015 Aug;166(1-3):334-8. doi: 10.1016/j.schres.2015.06.008. Epub 2015 Jun 24. PMID 26117157

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients transitioned from the acute phase study (D1050233 -NCT00790192) to the current study (D1050234) in a non-randomized fashion.
Groups:
- Lurasidone 80mg: Lurasidone 80mg/day in the acute phase study and flexibly-dosed lurasidone (40mg/day to 160mg/day) in the current study.
- Lurasidone 160 mg: Lurasidone 160mg/day in the acute phase study and flexibly-dosed lurasidone (40mg/day to 160mg/day) in the current study.
- Placebo-Lurasidone: Placebo in the acute phase study and flexibly-dosed lurasidone (40 mg/day to 160 mg/day) in the current study
- Quetiapine-Quetiapine: Quetiapine XR 600 mg/day in the acute phase study and flexibly-dosed quetiapine XR (200 mg/day to 800 mg/day) in the current study
Period: Overall Study
Arm/Group | Lurasidone 80mg | Lurasidone 160 mg | Placebo-Lurasidone | Quetiapine-Quetiapine
Started | 72 | 79 | 56 | 85
Completed | 32 | 46 | 29 | 33
Not Completed | 40 | 33 | 27 | 52
Not completed — Lack of Efficacy | 10 | 4 | 5 | 18
Not completed — Adverse Event | 5 | 5 | 3 | 4
Not completed — Lost to Follow-up | 5 | 5 | 2 | 9
Not completed — Protocol Violation | 6 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 14 | 15 | 12 | 19
Not completed — Administrative | 0 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 80mg | Lurasidone 160 mg | Placebo-Lurasidone | Quetiapine-Quetiapine | Total
Number analyzed (Participants) | 72 | 79 | 56 | 85 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (11.7) | 37.6 (11.7) | 37.5 (11.4) | 38.5 (10.4) | 37.6 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 27 | 21 | 33 | 97
  Male | 56 | 52 | 35 | 52 | 195
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 14 | 23 | 70
  Ukraine | 17 | 15 | 9 | 18 | 59
  Romania | 6 | 9 | 2 | 10 | 27
  Russian Federation | 11 | 15 | 12 | 17 | 55
  Colombia | 5 | 3 | 3 | 4 | 15
  India | 15 | 22 | 16 | 13 | 66

OUTCOME MEASURES:

1. Primary Outcome: Relapse of Psychotic Symptoms
Description: Time to relapse will be defined as the earliest occurrence of any of the following:
  * Worsening of >= 30% positive and negative syndrome scale total score from NCT00790192 and clinical global impression-severity sub-scale >=3
  * rehospitalization for worsening of psychosis
  * emergence of suicidal ideation, homicidal ideation and/or risk of harm to self or others Comparison of time to relapse of psychotic symptoms between lurasidone and quetiapine XR after 1 year as analyzed using the Cox proportional hazard model with country as a covariate.
Time Frame: 12 Months
Population: The population for relapse analyses is the relapse population which consists of those subjects who are enrolled in the present study, demonstrated response to 6 weeks of treatment with either lurasidone or quetiapine XR in study D1050233-NCT 00790192, and who took at least one dose of study medication in the present study.
Measure: Number; unit: participants
Groups:
- Lurasidone-Lurasidone: Lurasidone 80 mg/day or lurasidone 160 mg/day in the acute phase study and flexibly-dosed lurasidone (40 mg/day to 160 mg/day) in the current study.
Arm/Group | Lurasidone-Lurasidone | Quetiapine-Quetiapine
Number analyzed (Participants) | 139 | 79
participants | 29 | 21 [1 to 1]
Statistical Analysis 1: Comparison: Lurasidone-Lurasidone vs Quetiapine-Quetiapine; Comparison of time to relapse of psychotic symptoms between LUR-LUR and QXR-QXR as analyzed using the Cox proportional-hazards model; Test type: Non-Inferiority or Equivalence — This is a non-inferiority analysis. Lurasidone will be declared as effective as quetiapine XR in preventing relapse if the upper bound of a 2-sided 95% confidence limit for the hazard ration of lurasidone vs. quetiapine is no greater than an equivalence hazard ratio margin of 1.93; COX Proportional Hazards Model — There is no hypothesis tested. Since this was a non-inferiority study, the upper bound of the 95% CI for the hazard ratio was compared to the pre-specified margin of 1.93 to demonstrate the non-inferiority of lurasidone compared to Quetiapine XR; Hazard Ratio (HR) = 0.728, 95% CI 2-sided [0.410 to 1.295]

2. Secondary Outcome: Change From the Acute Phase Baseline to Month 6 of the Double-blind Treatment in the CogState Computerized Cognitive Scores.
Description: The battery has seven outcome measures that measure the cognitive constructs. The seven domains are: detection, identification, one back task, international shopping list task, one card learning task, Groton maze learning task and social emotional matching. The standardized scores for each subject at each assessment will then be averaged to yield a composite score. There are no maximum or minimum values, however a higher score indicates improved performance on the cognitive constructs. The change score is change from baseline to month 6.
Time Frame: Baseline and 6 Months
Population: The population is the intent to treat population which consists of those enrolled subjects who receive at least one dose of study medication and have either a PANSS or CGI-S baseline and post baseline measurements
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone-Lurasidone | Quetiapine-Quetiapine
Number analyzed (Participants) | 86 | 41
units on a scale | 0.22 [0.06 to 0.38] | -0.03 [-0.26 to 0.20]

3. Secondary Outcome: Change From the Acute Phase Baseline to the End (Month 12) of the Double-blind Treatment in the Positive and Negative Syndrome Scale (PANSS)
Description: The PANSS is an interview-based measure of psychopathology severity in adults with psychotic disorders. Thirty items are rated using a Likert scale, from 1 - 7. The PANSS total score is the sum of thirty items ranging from 30 to 210 (higher score representing a worsening in psychosis).
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone-Lurasidone | Quetiapine-Quetiapine
Number analyzed (Participants) | 132 | 72
units on a scale | -34.6 [-38.3 to -30.9] | -25.7 [-30.9 to -20.6]

4. Secondary Outcome: Change From the Acute Phase Baseline to the End (Month 12) of the Double-blind Treatment in the Clinical Global Impression Severity Scale (CGI-S) Scores
Description: The CGI-S is a clinician-rated assessment of the subject's current illness state on a scale ranging from 1-7, where a higher score is associated with greater illness severity.
Time Frame: Baseline and 12 months
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lurasidone-Lurasidone | Quetiapine-Quetiapine
Number analyzed (Participants) | 132 | 72
units on a scale | -1.9 [-2.1 to -1.7] | -1.6 [-1.9 to -1.4]

ADVERSE EVENTS:
Arm/Group | Lurasidone 80mg | Lurasidone 160 mg | Placebo-Lurasidone | Quetiapine-Quetiapine
Serious Adverse Events (participants affected / at risk) | 9/72 | 6/79 | 2/56 | 17/85
Other Adverse Events (participants affected / at risk) | 44/72 | 51/79 | 35/56 | 53/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80mg (N=72) | Lurasidone 160 mg (N=79) | Placebo-Lurasidone (N=56) | Quetiapine-Quetiapine (N=85)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skeletal Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 6 (6)
Schizophrenia (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 9 (9)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Behavior (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 80mg (N=72) | Lurasidone 160 mg (N=79) | Placebo-Lurasidone (N=56) | Quetiapine-Quetiapine (N=85)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 6 (6) | 2 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (5)
Vomiting (Gastrointestinal disorders) | 3 (8) | 3 (4) | 3 (4) | 4 (7)
Weight Increased (Investigations) | 3 (6) | 6 (6) | 1 (1) | 7 (8)
Akathisia (Nervous system disorders) | 11 (16) | 8 (9) | 6 (9) | 2 (3)
Dystonia (Nervous system disorders) | 4 (7) | 1 (1) | 2 (6) | 1 (1)
Headache (Nervous system disorders) | 5 (7) | 11 (16) | 3 (5) | 8 (11)
Parkinsonism (Nervous system disorders) | 3 (5) | 6 (7) | 9 (12) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (6) | 2 (3) | 3 (4)
Insomnia (Psychiatric disorders) | 5 (5) | 7 (8) | 4 (4) | 8 (9)
Schizophrenia (Psychiatric disorders) | 5 (6) | 2 (2) | 2 (2) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.